CLINICAL TRIAL: NCT06496230
Title: EMPWR Pilot Trial: Treatment Retention in Medication for Opioid Use Disorder Among Pregnant and Postpartum Women
Brief Title: Open Trial of Technology-Enhanced Behavioral Intervention for Buprenorphine Retention in Pregnant and Postpartum People
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sara Witcraft, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00137982; K12DA031794 (NIH)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Pregnancy Related
Keywords: Anxiety; Mental Health; Pregnancy; Psychiatry; Sleep Disorders; Substance Use; Women's Health
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Psychological Well-Being; Sleep Wake Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empowering Pregnant Women and People Receiving Medications for Opioid Use Disorder (Experimental): EMPWR is a two-pronged intervention model comprised of 1) a provider-driven, telemedicine-based behavioral intervention to mitigate anxiety sensitivity and sleep deficiency and enhance peripartum buprenorphine retention, and 2) an adjunctive mobile application to promote patients' buprenorphine adherence and use of therapy skills learned through the behavioral intervention. The EMPWR therapy protocol is comprised of five 30-60-minute sessions delivered weekly or biweekly by a therapist during the second and/or third trimester of pregnancy, and three 30-minute booster sessions delivered months 1-3 postpartum.
  Interventions: Behavioral: Empowering Pregnant Women and People Receiving Medications for Opioid Use Disorder

INTERVENTIONS:
Behavioral: Empowering Pregnant Women and People Receiving Medications for Opioid Use Disorder — Two-pronged intervention model: 1) behavioral intervention utilizing interoceptive exposures and cognitive behavioral therapy for insomnia and, 2) mobile application that facilitates medication adherence.
  Other Names: EMPWR

SUMMARY:
This study involves testing how useful a technology-enhanced intervention is for pregnant people prescribed buprenorphine for the management of opioid use disorder. The intervention being studied is a brief therapy protocol and a mobile application. Participation involves four 60-minute therapy appointments during pregnancy, and four 30-minute therapy appointments at the end of pregnancy through 3 months postpartum. The mobile application will be accessible for at least the duration of the study. Participants will also be asked to complete questionnaires at enrollment and again at 1-month postpartum and 3-months postpartum, will send monthly photos of their prescription bottle/box, and will be contacted randomly throughout the study to perform a medication count. The total duration of the study is between 5-9 months depending on when you enroll (early second trimester-mid third trimester). Compensation is provided.

DETAILED DESCRIPTION:
Medication for opioid use disorder (MOUD) can effectively prevent overdose and death for pregnant and postpartum people with opioid use disorder (OUD). Yet, only half of birthing people continue to use MOUD postpartum, increasing risk for overdose two-fold. This study will evaluate acceptability of a technology-enhanced behavioral intervention that aims to improve retention in and adherence to MOUD during the peripartum period. The intervention contains a brief behavioral intervention targeting malleable risk factors for treatment dropout, opioid cravings, and return to illicit opioid use: anxiety sensitivity and sleep deficiency. An adjunctive mobile application will supplement therapy sessions and contains a medication adherence feature involving daily (or multiple/day) notification reminder to take medication at a scheduled time and dose consistent with the participant's prescription.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant and less than 33 weeks gestational age,
* History of OUD within past 3 years,
* Confirmed prescription for sublingual buprenorphine products (i.e., Suboxone, Subutex, Zubsolv) for the purpose of treating OUD,
* Living in the United States,
* Between 18-45 years of age.

Exclusion Criteria:

* Carrying multiples (i.e., twins, triplets, etc.);
* High-risk pregnancies including the following conditions: hyperemesis defined as hospitalization for intractable nausea and vomiting, hypertensive disorders of pregnancy (e.g., gestational hypertension, preeclampsia), placenta previa, or vaginal bleeding in current pregnancy after the first trimester;
* Current psychotic symptoms and/or active suicidal intent;
* Experiencing cognitive or emotional impairment that precludes providing informed consent;
* Incarcerated/pending incarceration or institutionalized during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 26 pregnant individuals will be recruited to participate in this study.
Enrollment: 26 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 1 year
  Feasibility of the intervention (e.g., Recruitment: 20 pregnant women with OUD prescribed buprenorphine; Study retention: ≥50% participants retained through 3-month postpartum assessment; Protocol adherence: ≥50% attend all EMPWR therapy sessions;145 Satisfaction: qualitative feedback to assess what participants liked/did not like about the intervention)

SECONDARY OUTCOMES:
Buprenorphine retention | 6 months
  Prescription drug monitoring program (y/n)
Buprenorphine adherence | 6 months
  Mobile application data, medication possession ratios (%)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Witcraft, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No